CLINICAL TRIAL: NCT00871312
Title: A Randomized, Double-blinded, Parallel Group, Placebo-Controlled, Multi-Center Trial of Topical Wound Oxygen Therapy in the Treatment of Diabetic Lower Extremity Ulcers
Brief Title: Evaluation of Topical Wound Oxygen (two2) Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate meaning unable to complete the study in a timely manner
Sponsor: AOTI Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOTI-001
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Diabetic Ulcer
Keywords: diabetes; diabetic; wound; ulcer; lower extremity; foot; oxygen; hyperbaric; topical wound oxygen
MeSH Terms: conditions — Diabetes Mellitus; Wounds and Injuries; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Wound Oxygen Therapy (Active Comparator): Subjects will receive four 90 minute treatments of two2 therapy per week
  Interventions: Device: Topical wound oxygen therapy
- Placebo Therapy (Placebo Comparator): Subjects will receive four 90 minute treatments of Placebo two2 therapy per week
  Interventions: Device: Topical wound oxygen Placebo

INTERVENTIONS:
Device: Topical wound oxygen therapy — 90 minutes 4 days per week Active Topical Oxygen Therapy
  Arms: Topical Wound Oxygen Therapy
Device: Topical wound oxygen Placebo — 90 mins per day 4 days per week Placebo Therapy
  Arms: Placebo Therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Topical Wound Oxygen (two2) therapy system on the healing of diabetic lower extremity ulcers.

DETAILED DESCRIPTION:
The AOTI two2 therapy trial is a randomized, double-blinded, parallel group, placebo-controlled, multi-center study intended to evaluate the efficacy of Topical Wound Oxygen (two2) therapy in relation to placebo when added to standard of care in the treatment of diabetic lower extremity ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal representative has read, understands, and has signed the Institutional Review Board (IRB)-approved Informed COnsent Form (ICF) prior to enrollment in the study;
* Subject is 18 years of age or older;
* Subject has a current diagnosis of Type I or Type II diabetes mellitus;
* Subject has a diabetic lower extremity ulcer;
* Subject's index ulcer is at least 1.0cm2 in area;
* Subject's index ulcer is a superficial, partial or full thickness skin ulcer (Wagner Classification System I, II or III) which has been present for at least 4 weeks at the time of initial screening that has not improved with standard of care;
* Subject's index ulcer appears to be free of sinus tracts and tunneling;
* Subject's index ulcer exhibits no signs of moderate or severe clinical infection;
* In the event of multiple wounds on the same foot, the index ulcer will be the largest ulcer meeting the other inclusion criteria;
* In the event of multiple wounds on the same foor, the index ulcer is at least 2 cm from any additional wound edge;
* Women of childbearing potential must not be pregnant or lactating;
* Subject and/or caregiver are willing and able to comply with all specified care and visit requirements, and subject has a reasonable expectation of completing the study;
* Subject must be fit to undertake the study trial in the opinion of the referring doctor
* Subject's Great Toe pressure is greater than 20mmHg.

Exclusion Criteria:

* Subject is currently enrolled in another investigational device or drug trial, or has been previously enrolled in investigative research for a device or pharmaceutical agent within the last 30 days;
* Subject's index ulcer has gangrene or gangrene is located on any part of the foot with the index ulcer;
* Subject has an acute and/or active Deep Vein Thrombosis;
* Subject is currently receiving or has received in the last six (6) months radiation or chemotherapy;
* Subject has received growth factor therapy within seven (7) days prior to initial screening;
* Subject has a significant medical condition that would impair wound healing, for example: severe liver disease, aplastic anemia, scleroderma, malnutrition, malignancy, etc;
* Subject has known or suspected osteomyelitis;
* Other than debridement, the underlying wound pathology requires surgical correction for the index ulcer to heal;
* Subject is receiving or has received corticosteroids (all applications), immunosuppressive agents, or other drugs that would impair wound healing within seven (7) days prior to initial screening or is anticipated to require them during the course of the study;
* Subject has an acute or active Charcot foot per clinical and radiology results or significant bony prominences that would preclude adequate off-loading with the standard off-loading device. The presence of Charcot foot in itself does not exclude the subject;
* Subject has known HIV, hepatitis, active cancer (except basal cell and non-melanoma skin cancer), or a bleeding disorder;
* Subject is undergoing renal dialysis;
* Subject suffers from known alcohol or drug abuse;
* Use of the standard off-loading device is contra-indicated or cannot be appropriately fitted to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Wound closure | 12 Weeks

SECONDARY OUTCOMES:
The time to wound closure | Variable
The degree of wound closure | 4, 8, and 12 weeks
The percentage of tissue types | 4, 8 and 12 weeks
The type and amount of wound drainage or exudates | 4, 8 and 12 weeks
The level of wound pain | 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Edsberg, Ph.D., Principal Investigator — Daamen College
Locations (3):
- AOTI Clinic, Buffalo, New York, United States
- Canada (2):
  - Community Dermatology & Wound Healing Clinic, Mississauga, Ontario
  - Wound Care Clinic, Saint Catherines, Ontario